CLINICAL TRIAL: NCT00790452
Title: A Randomized Phase II Trial of Aspirin for Primary Prophylaxis of Venous Thromboembolism in Glioblastoma
Brief Title: Aspirin Prophylaxis for Venous Thromboembolism in Glioblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007-0266
Record Dates: First submitted 2008-11-07; First posted 2008-11-13 (Estimated); Results first posted 2011-12-08 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-11

CONDITIONS: Glioblastoma
Keywords: Brain; Hematologic Disorder; Venous Thromboembolism; Glioblastoma; Aspirin; Placebo; VTE; ASA; DVT
MeSH Terms: conditions — Glioblastoma; Hematologic Diseases; Venous Thromboembolism | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Aspirin) (Active Comparator): Aspirin 325 mg/day orally
  Interventions: Drug: Aspirin
- Group 2 (Placebo) (Placebo Comparator): Tablet/day orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — 325 mg daily by mouth
  Other Names: ASA
  Arms: Group 1 (Aspirin)
Drug: Placebo — Tablet daily by mouth
  Arms: Group 2 (Placebo)

SUMMARY:
Primary objective:

To determine whether aspirin (ASA) can lower the incidence of Venous Thromboembolism(VTE) in patients with Glioblastoma (GBM).

Secondary objectives:

To determine clinical and laboratory factors which are associated with increased risk of VTE

If it is determined that ASA reduces the incidence of VTE in patients with GBM, then to determine the clinical and laboratory factors which are associated with an increased benefit from the drug.

DETAILED DESCRIPTION:
Study Drug:

Aspirin is designed to make blood less "sticky" and reduce its chances of clotting. By making blood less sticky, it may be less likely to allow a clot to form.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to 1 of 2 study groups. If you are assigned to Group 1, you will take aspirin. If you are in Group 2, you will take a placebo. A placebo is a substance that looks like the study drug but has no active ingredients. You will have an equal chance of being placed in either group. Neither you nor your study doctor will know what group you are in. In case of an emergency, the study staff will be able to find out which group you are in.

Study Drug Administration:

If you are assigned to Group 1, you will take 1 aspirin tablet, once a day, by mouth. Aspirin should be taken with food and may be taken at any time during the day.

If you are assigned to Group 2, you will take 1 placebo tablet once a day, by mouth. The placebo should be taken with food and may be taken at any time during the day.

Study Visits:

While on study you will have tests and procedures performed at the same time as each routine clinical visit and when the study doctor thinks it may be necessary. The following tests and procedures will be performed:

* You will have a physical exam.
* You will be checked for VTE at each visit.
* Blood (2 teaspoons) will be drawn for routine tests at least once every 8 weeks. Blood samples will not be routinely collected if you are not receiving any chemotherapy.
* Blood (about 1 teaspoon) will be drawn to see how well your blood clots about 4 months after you begin treatment. If you show signs of VTE, this test will be done on the first visit after the signs are shown.

Length of Study:

You may remain on-study for as long as you are benefiting. If the disease gets worse or intolerable side effects occur, you may be taken off of the study.

End of Study Visit:

Once you are off-study, you will have an end-of-study visit. At this visit, the following tests and procedures will be performed:

* Your complete medical history will be recorded.
* You will have a physical exam.
* You will have performance status evaluation.
* You will be asked about any medications you may be taking.
* You will be checked for VTE.
* Blood (about 1 teaspoon) will be drawn to see how well your blood clots.
* If you have symptoms of VTE, you will have a Doppler ultrasound test of your legs.

Follow-up:

The study staff will call you or a member of your family every 3 months, after your last clinic visit, to follow your health status.

This is an investigational study. Aspirin is approved by the FDA and commercially available. Its use in lowering the risk of VTE is investigational. Aspirin, and the study-related tests/procedures will be provided free of charge to you while on this study. Up to 224 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven supratentorial malignant WHO grade IV gliomas will be eligible for this protocol. These include glioblastoma multiforme (GBM) and gliosarcoma.
2. The patient must have contrast enhancement documented on MRI or CT associated report.
3. Understand and voluntarily sign an informed consent form.
4. Karnofsky performance status of 60 or greater at study entry.
5. Able to adhere to the study visit schedule and other protocol requirements.
6. No more than 16 weeks from the diagnosis of glioblastoma, which is defined as the date of the surgical procedure establishing the histologic diagnosis operation.
7. No more than 1 recurrence of tumor following initial diagnosis.
8. Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply: 1). At least 1 week has elapsed since the operation. 2). Any blood products visible on brain imaging (CT or MRI) are documented by the treating clinician or radiology report as residual and not active bleeding.
9. Laboratory test results within these ranges: 1). The following two laboratory studies should be performed within14 days from enrollment if receiving cytotoxic chemotherapy; </= 90 days otherwise. (a) Platelet count greater than or equal to 50 x 10^9/L. (b). Hematocrit greater than or equal to 29.0.
10. (10. continued) 2) For the following two laboratory studies, any documented prior normal value is acceptable (including outside institution results) provided that the patient is not taking anticoagulants such as coumadin. If not available, they should be checked. (a) Creatinine less than or equal to 1.5. (b) International Normalized Ratio less than or equal to 1.3. 3) D-Dimer blood test within the institutional normal level within 7-days of study entry
11. Age 18 years or greater at the time of signing the informed consent form. Background data regarding VTE is from adults and may not be applicable to children.
12. This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Patients will be recruited with no preference to gender.

Exclusion Criteria:

1. Patient is unable to provide informed consent.
2. Pregnant or lactating females, as aspirin may impart addition risk for this patient population.
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study as determined by the enrolling physician.
4. Known hypersensitivity or allergy to aspirin.
5. Clinical indication or use of agents with potential of increased bleeding risk via alteration of coagulation pathways or platelet activation including (but not limited to) warfarin, heparins, aspirin, dipyridamole, celecoxib, NSAIDs and clopidogrel. (1) Any use of warfarin, heparinoids, dipyridamole, clopidogrel for greater than 2 consecutive weeks in the prior 6 months (2) Occasional use of NSAIDs, aspirin, or COX-2 inhibitors is not an exclusion if taken on an "as needed" basis less than once per week on average.
6. Diagnosed or suspected peptic ulceration within the last 5 years
7. History of gastrointestinal bleeding within the last 5 years.
8. History of major bleeding (NCIC grade 3-4) within the last 5 years.
9. Hereditary coagulopathy or hypercoagulable state.
10. Anticipated refusal of blood products or maximal supportive care
11. History of spontaneous (non-surgical) intracranial hemorrhage during lifetime.
12. Active or recent uncontrolled gastrointestinal symptoms such as nausea, vomiting, and diarrhea, which are unresolved or within 2 weeks of resolution, or are anticipated to recur.
13. Patient who would be unlikely or unwilling to follow-up at MD Anderson at or more frequently than every 3 months.
14. No exclusion to this study will be based on race. Minorities will actively be recruited to participate. The malignant glioma patient population treated at MDACC over the past year is as follows: American Indian or Alaskan Native - 0. Asian or Pacific Islander - <2%. Black, not of Hispanic Origin - 3%. Hispanic - 6%. White, not of Hispanic Origin - 88%. Other or Unknown - 2%. Total-100%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor A Levin, MD,BS, Principal Investigator — The University of Texas MD Anderson Cancer
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 28, 2008 to October 26, 2009. All patient recruitment attempted to UT MD Anderson Cancer Center.
Pre-assignment Details: The only participant enrolled was removed from the study due to a drug supply issue, and the study terminated early.
Period: Overall Study
Arm/Group | Group 1 (Aspirin) | Group 2 (Placebo)
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Drug supply issue | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Aspirin) | Group 2 (Placebo) | Total
Number analyzed (Participants) | 1 | 0 | 1
Age Continuous [Median (Full Range); unit: years] | 53 [53 to 53] |  | 53 [53 to 53]
Gender [Number; unit: participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Frequency of VTE Events
Description: Occurrences of Venous Thromboembolism (VTE) events in each study arm of a randomized placebo controlled trial of aspirin in GBM Patients.
Time Frame: VTE evaluation with study visits (4 weeks) for up to 2 years
Population: Analysis was to be per protocol, study terminated early with no analysis. Only enrolled participant to the study was prematurely taken off the study due to a drug supply issue.
Measure: Number; unit: participants
Arm/Group | Group 1 (Aspirin) | Group 2 (Placebo)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Group 1 (Aspirin) | Group 2 (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
Study terminated early due due to a drug supply issue.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No